CLINICAL TRIAL: NCT00497406
Title: A Pilot Study to Evaluate the Feasibility of Combining Submandibular Salivary Gland Transfer Procedure and Intensity Modulated Radiation Therapy (Helical Tomotherapy) to Reduce Dryness of Mouth (Xerostomia) in Head and Neck Cancer Patients After Surgery
Brief Title: A Pilot Study to Evaluate the Feasibility of Combining Submandibular Salivary Gland Tx & IMRT Tomo to Reduce Xerostomia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HN-4-0027/ethics 22128
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
Keywords: submandibular salivary gland transfer; intensity-modulated radiation therapy; helical tomotherapy; reduction of xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Salivary gland transfer — Retrograde flow method
Procedure: Helical Tomotherapy treatment — total of 30 fractions

SUMMARY:
A study for head and neck cancer patients to evaluate the feasibility of combining salivary gland transfer surgical procedure and IMRT helical tomotherapy to reduce dryness of mouth.

DETAILED DESCRIPTION:
Background Information Radiation therapy is used in a definitive manner or as an adjunct to surgery in most of the head and neck cancer patients which inevitably lead to xerostomia (salivary gland dysfunction) in almost all patients. Xerostomia is debilitating condition which adversely affects the deglutition, mastication, gustation, speech and lead to increased susceptibility of structures in mouth to infection. Xerostomia may also interfere with nutrition and sleep of patient and thereby has a significant negative impact on patient's quality of life. Various modalities have been explored to prevent or decrease the incidence of xerostomia and the most successful methods are; use of Intensity modulated radiotherapy (IMRT) to spare the parotid salivary gland from radiation, Sparing submandibular salivary gland from radiation by it's transfer to sub mental space, use of Amifostine to protect salivary glands from radiation and use of cholinergic agonists like pilocarpine to stimulate salivary secretion. Both amifostine and pilocarpine are associated with significant side effects and amifostine is too costly to be used in routine practice. At our center, we were successful in decreasing the incidence of xerostomia significantly by using either IMRT sparing parotid gland (Parliament et al 2004) or submandibular gland transfer (SGT) sparing submandibular gland (Jha et al 2003)without compromising the tumor control rates. Both these modalities were not associated with any added toxicity which makes these methods superior to pilocarpine and amifostine. To improve upon our results by sparing both the major salivary glands, we plan to explore a combined approach of IMRT and SGT in head and neck cancer patients after surgery. For IMRT we had used "step-and-shoot" technique on a Varian 2300 EX linac with 120-leaf Millenium MLC. Since December 2002, the Cross Cancer Institute has had a helical tomotherapy unit at its disposal for IMRT and a planning study (van Vulpen et al 2005) conducted comparing the step-and-shoot IMRT and Helical tomotherapy for 5 oropharynx patients showed that tomotherapy plans compared favorably with step- and-shoot plans regarding sparing of the parotid glands. Hence we intend to use helical tomotherapy as an IMRT tool for this study.

Objectives - primary and secondary Primary objective is to assess the feasibility of sparing parotid and transferred submandibular gland by combining IMRT using helical tomotherapy with SGT in cancers of oropharynx, larynx, hypopharynx after primary surgery and patients with unknown primary cancer with neck nodes after neck dissection.

Secondary objectives are to assess the incidence of xerostomia subjectively by xerostomia specific &University of Washington Quality of Life Head and Neck Symptom questionnaire and objectively by sialometry and salivary scintigraphy after parotid-sparing IMRT+ SGT. We also intend to evaluate the speech and swallowing function of patients before and after radiation. All these functional outcomes will be correlated with the dose-volume histograms of salivary glands.

Study Design Primary squamous cell carcinomas of oropharynx, larynx, hypopharynx Unknown primary with neck nodes with squamous cell carcinoma histology

? Radical surgery for primary cancers of oropharynx, larynx, hypo pharynx or Neck dissection for unknown primary with neck nodes

+ Selective neck dissection(level I-III) and SGT on opposite side for lateralized primary and on the side of N0 neck for midline primary

?

IMRT with Helical tomotherapy sparing the parotid glands and transferred submandibular gland + chemotherapy

Statistical Analysis - Power and/or Sample Size Relation This pilot study on 12 patients will be considered as feasible if we can limit the mean radiation dose to one parotid and one transferred submandibular gland to less than 26Gy while giving a radiation dose of 60Gy to PTV 1 and 54 Gy to PTV 2 .We intend to report only the descriptive statistics related to incidence and severity of xerostomia.

Stopping Rules Radiation treatment will be withheld if any patient develops acute toxicity of RTOG grade?4 or any unpredictable adverse events. Other than this, the decision to stop/delay treatment if clinically indicated will be at the discretion of the treating physician.

Data Safety Monitoring Committee Data will be handled by Juliette Jordan as per rules of Alberta Cancer Board. Recruitment & Eligibility Criteria " Twelve patients with histologically proven newly diagnosed squamous cell carcinoma of the oropharynx, larynx, hypo pharynx and unknown primary cancer with neck nodes after primary surgery will be recruited to this study.

" AJCC stage I-IV patients are eligible provided they are M0 and N0-2b. " age 18, and Karnofsky performance status 70 " patients must sign a study-specific informed consent form " Patients with: N3/N2C/ M1 disease, salivary gland diseases like Sjogren's syndrome, prior or concurrent malignancy, prior or concurrent malignancy, pre-epiglottic space involvement on pathological examination, involvement of level I nodes on either side of neck, post op recurrent disease at presentation will not be eligible for this study.

Additional procedures and investigations that will be done in this study are outlined below.

Submandibular Gland Transfer We are using the retrograde flow method for gland transfer. Retrograde flow flaps are well established techniques that are extensively used in finger and hand reconstructions. The gland is dissected and left pedicled on the artery, vein, and submandibular region. The great auricular nerve is dissected, harvested and preserved for later use. The facial artery and vein are cut just proximal to their branches supplying the gland. The efferent nerves of the submandibular ganglion are also cut. The gland is then repositioned in the submental space after the mylohyoid muscle is cut to allow the repositioning of the submandibular duct. The efferent nerves of the submandibular region are then reattached to the gland with the greater auricular nerve interposition graft. In our experience (more than 200 patients so far) we have experienced only one case of recurrence of tumor in the grafted area.

Sialometry Whole salivary flow rates, unstimulated and stimulated, will be measured from the floor of the mouth and labial vestibule preoperatively and at 2-3 weeks after surgery before start of radiation treatment. After radiation treatment, flow evaluation will be done at 6 months and 12 months. Each time, the flow rate will be measured at rest and after stimulation. Stimulated flow rates will be measured by dropping 0.2 ml of 6% citric acid solution on the dorsal surface of the tongue every 30 seconds (Dawes 1975).Salivary samples will be collected by means of a an appliance (Pederson et al 1985) consisting of a Drummond micropipette holder (for use with 20 microlitre micropipettes) fitted with a 2 ml latex dropper bulb. A 2.5 cm length of 50 microlitre micropipette is inserted into the holder until its outer end no longer protrudes. During collection, the patient tips the head slight forward to produce pooling of saliva at the anterior floor of mouth and mandibular labial vestibule. The micropipette extruding from the end of the collection device is used to aspirate the pooled salivary secretions from these two sites. As saliva flows up the micropipette, it spills into the glass sleeve of the collection device between the top of the silicon end-piece and the top of the micropipette.

Salivary Scintigraphy Salivary gland scintigraphy will be carried out using sodium pertechnate 99mTc 04,before surgery,2-3 weeks after surgery and 6 months,12 months after radiation therapy to evaluate the morphology and function of the "transferred gland". This will be compared with the salivary gland morphology and function that will receive radiation treatment. After 148 MBq of 99mTc 04 is rapidly injected with computer acquisition of 1 min frames, for a total of 30 min. After 15 minutes time point, the patient is requested to suck on the juice of a lemon by a straw, in order to provoke salivary secretion.

Speech and Swallowing Assessments This assessment will be done at the Head and neck Surgery Functional Assessment Laboratory is housed within COMPRU at the Misericordia Hospital. Each patient will be scheduled for 4 predetermined assessment visits:1) preoperative; 2) 2-4 weeks postoperative; 3) 6-months post-radiation therapy; and 4) 1-year post radiation therapy. At each of these sessions, speech, mastication, deglutition, and quality of life will be assessed. Speech function will be assessed by recording the voice of patient using audiotapes. Masticatory efficiency will be assessed using an electrognathograph (BioPak, Version 2.0, Milwaukee, WI), a clinical tool that measures mandibular movement using a sensory array to track the position of a magnet placed on a patient's mandibular incisors. After placement of both the magnet on the mandibular dentition and the sensory array on the head, each patient will be asked to chew a wine gum and ¼ of a digestive cookie. Various aspects of mastication will be assessed including the number of chewing strokes and time passing before the first swallow of both the candy and the cookie. Swallowing function will be assessed by fluoroscopic visualization while the patient is swallowing food substances of different consistencies coated with Barium.

ELIGIBILITY:
Inclusion Criteria:

* histologically-proven newly-diagnosed squamous cell carcinoma of oropharynx, larynx, hypopharynx and unknown primary of cancer with neck node metastasis after primary surgery
* AJCC stage I-IV patients are eligible provided they are MO and NO-2b
* 18 years of age or older
* KPS of 70 or greater

Exclusion Criteria:

* N3/N2C disease or M1 disease
* salivary gland disease i.e. Sjogren's syndrome
* prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for at least 5 years
* prior radiotherapy to the head and neck region
* lymph node involvement (level I-III) or proximity of disease to submandibular gland on the side chosen for salivary gland transfer on frozen section or permanent pathological evaluation
* pre-epiglottic space involvement on pathological examination
* involvement of level I nodes on either side of neck
* post-op recurrent disease at presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-12; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
reduction of Xerostomia after surgery | 2-3 weeks after surgery, 6 months and 12 months
  combining submandibular salivary gland transfer procedure and intensity modulated radiation therapy (helical tomotherapy) to reduce dryness of mouth in head and neck cancer patients after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rufus Scrimger, MD, FRCPC, Study Chair — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada